CLINICAL TRIAL: NCT03759847
Title: Fluid Intake App for Management of Volume Intake in Patients Receiving Chronic Hemodialysis Therapy
Brief Title: Development of Fluid Intake App for Management of Fluid Intake During Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00048561
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-02

CONDITIONS: Weight Gain
Keywords: hemodialysis; fluid intake; Interdialytic weight gain
MeSH Terms: conditions — Weight Gain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Comparison of interdialytic weight gain with fluid intake as recorded by fluid app
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vanguard (Experimental): Participants in this arm will use the fluid intake app and take a survey to test the fluid intake monitoring app for both safety and design issues.
  Interventions: Other: Fluid intake app; Other: Survey

INTERVENTIONS:
Other: Fluid intake app — Use of fluid app to monitor intake of fluids
Other: Survey — A survey will be used to assess the usability of the app (ease of use in general, ease of capturing fluid intake data, including the choice of pre-selected volumes for fluid containers, reasons for not using the app more frequently, the usefulness of the app notifications, ease of sending data to the study coordinator for review) as well as to collect recommendations for changes to the app itself.

SUMMARY:
Methods are needed to help decrease interdialytic weight gains in hemodialysis patients. One potential method for accomplishing this goal is to develop an app for smartphones that allow patients to track their fluid intake throughout the course of the day. This protocol is designed to test the safety and efficacy of this app, followed by use of the app in patients with large fluid weight gains between HD sessions. In the Vanguard phase, patients without large interdialytic fluid gains (less than 4%) will use the app to to determine the association between the interdialytic weight gain and the fluid consumed as recorded by use of the app for each interdialytic period. The app will be modified, if needed, prior to initiation of the full scale trial.

DETAILED DESCRIPTION:
For the Vanguard phase of the trial, a survey will be used to assess the usability of the app as well as to collect recommendations for changes to the app itself (appendix one). For this Vanguard phase study, the survey for participants will be designed to assess the usability of the app (ease of use in general, ease of capturing fluid intake data, including the choice of preselected volumes for fluid containers, reasons for not using the app more frequently, the usefulness of the app notifications, ease of sending data to the study coordinator for review). The survey for the study coordinator will be designed to assess the ease of reviewing data from participants and the perceived difficulty of patient use of the app.

ELIGIBILITY:
Inclusion Criteria:

* Subject, upon briefing of the content of the present study, fully understanding and agreeing to its objective and having given written (dated and signed) informed consent form to take part in the study.
* Adult chronic hemodialysis patients who are at least 18 years of age
* Average interdialytic fluid gains of less than 4% of body weight for both weekdays and weekends for a 30 day period
* Access to a smartphone for use of the app and comfort with using apps on a regular basis
* Access to a smartphone running under either iOS or Android operating systems
* Sufficient knowledge and understanding of the English language to use the application available only in English (US) language
* Mental capacity to use and understand the fluid management app
* Willingness to share intake data collected with the research team

Exclusion Criteria:

* Scheduled for a living related renal transplant in the next four months
* Class III or IV heart failure
* Need for chronic oxygen therapy due to pulmonary disease
* Hospitalization within 30 days of entry into the study
* Current participation in a randomized clinical trial or in the exclusion period of another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Amount of interdialytic weight gain | 1 month
  The amount of weight gain as recorded by use of the app for each interdialytic period. The association between the interdialytic weight gain and the fluid consumed will be assessed by a repeated measures analysis of variance with an unstructured covariance matrix.
Amount of fluid consumed | 1 month
  The fluid consumed as recorded by use of the app for each interdialytic period. The association between the interdialytic weight gain and the fluid consumed will be assessed by a repeated measures analysis of variance with an unstructured covariance matrix.

SECONDARY OUTCOMES:
Number of patients who experienced a 50% increase in fluid intake during app use | 1 month
  This will be a safety evaluation to ensure that no participants had more than a 50% increase in fluid intake while using the app. It will be described using descriptive statistics.
Number of days that the app was used | 1 month
  This will be the determination of the number of days that the app was used.
Number of days that the app was used by day of the week | 1 month
  Differences in app use by specific days of the week. This is a sub analysis using days of the week.
Number of days that the app was used by dialysis or non-dialysis days | 1 month
  Differences in app use by specific days of the week, including dialysis and non-dialysis days. This is a sub analysis using dialysis versus non-dialysis days.
Ratio of weight of liquid intake | 1 month
  Agreement between fluid intake and weight gain will be described using descriptive statistics by the ratio of weight of liquid intake between two visits over the interdialytic weight gain

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rocco, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Kidney Foundation. KDOQI Clinical Practice Guideline for Hemodialysis Adequacy: 2015 update. Am J Kidney Dis. 2015 Nov;66(5):884-930. doi: 10.1053/j.ajkd.2015.07.015. PMID 26498416
- [Background] United States Renal Data System. National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases, Bethesda, MD
- [Background] Eknoyan G, Beck GJ, Cheung AK, Daugirdas JT, Greene T, Kusek JW, Allon M, Bailey J, Delmez JA, Depner TA, Dwyer JT, Levey AS, Levin NW, Milford E, Ornt DB, Rocco MV, Schulman G, Schwab SJ, Teehan BP, Toto R; Hemodialysis (HEMO) Study Group. Effect of dialysis dose and membrane flux in maintenance hemodialysis. N Engl J Med. 2002 Dec 19;347(25):2010-9. doi: 10.1056/NEJMoa021583. PMID 12490682
- [Background] FHN Trial Group; Chertow GM, Levin NW, Beck GJ, Depner TA, Eggers PW, Gassman JJ, Gorodetskaya I, Greene T, James S, Larive B, Lindsay RM, Mehta RL, Miller B, Ornt DB, Rajagopalan S, Rastogi A, Rocco MV, Schiller B, Sergeyeva O, Schulman G, Ting GO, Unruh ML, Star RA, Kliger AS. In-center hemodialysis six times per week versus three times per week. N Engl J Med. 2010 Dec 9;363(24):2287-300. doi: 10.1056/NEJMoa1001593. Epub 2010 Nov 20. PMID 21091062
- [Background] Chan CT, Greene T, Chertow GM, Kliger AS, Stokes JB, Beck GJ, Daugirdas JT, Kotanko P, Larive B, Levin NW, Mehta RL, Rocco M, Sanz J, Schiller BM, Yang PC, Rajagopalan S; Frequent Hemodialysis Network (FHN) Trial Group. Determinants of left ventricular mass in patients on hemodialysis: Frequent Hemodialysis Network (FHN) Trials. Circ Cardiovasc Imaging. 2012 Mar;5(2):251-61. doi: 10.1161/CIRCIMAGING.111.969923. Epub 2012 Feb 23. PMID 22360996
- [Background] Chan CT, Greene T, Chertow GM, Kliger AS, Stokes JB, Beck GJ, Daugirdas JT, Kotanko P, Larive B, Levin NW, Mehta RL, Rocco M, Sanz J, Yang PC, Rajagopalan S; Frequent Hemodialysis Network Trial Group. Effects of frequent hemodialysis on ventricular volumes and left ventricular remodeling. Clin J Am Soc Nephrol. 2013 Dec;8(12):2106-16. doi: 10.2215/CJN.03280313. Epub 2013 Aug 22. PMID 23970131
- [Background] Assimon MM, Wenger JB, Wang L, Flythe JE. Ultrafiltration Rate and Mortality in Maintenance Hemodialysis Patients. Am J Kidney Dis. 2016 Dec;68(6):911-922. doi: 10.1053/j.ajkd.2016.06.020. Epub 2016 Aug 26. PMID 27575009
- [Derived] Rocco MV, Rigaud M, Ertel C, Russell G, Zemdegs J, Vecchio M. Fluid Intake Management in Maintenance Hemodialysis Using a Smartphone-Based Application: A Pilot Study. Kidney Med. 2023 Jul 26;5(9):100703. doi: 10.1016/j.xkme.2023.100703. eCollection 2023 Sep. PMID 37663954

DOCUMENTS (1):
  • Informed Consent Form (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT03759847/ICF_000.pdf